CLINICAL TRIAL: NCT02568566
Title: A Prospective, Single-arm, Open-label, Non-randomized, Phase IIA Trial of a Nonavalent Prophylactic HPV Vaccine to Assess Immunogenicity of a Prime and Deferred-booster Dosing Schedule Among 9-11 Year-old Girls and Boys
Brief Title: Recombinant Human Papillomavirus Nonavalent Vaccine in Preventing Human Papilloma Virus in Younger Healthy Participants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2015-01645; NCI-2015-01645 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01CN00031 (NIH); N01-CN-2012-00031; 1512261519 (Other: Banner University Medical Center - Tucson); UAZ2015-05-01 (Other: DCP); P30CA023074 (NIH)
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (Gardasil 9) (Experimental): Patients receive recombinant human papillomavirus nonavalent vaccine IM at baseline (priming injection) and at 24 and 30 months (booster injections).
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine

SUMMARY:
Human papillomavirus (HPV) is a common sexually-transmitted virus which causes infections that usually last only a few months, but sometimes can last a long time and cause cancers of the cervix, vagina, vulva, anus or oropharynx over many years among adults. This phase IIA trial studies how well does the nonavalent HPV vaccine (which can prevent nine different types of HPV) work when given in an alternative dosing schedule to heathy young research participants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the persistence and stability of serologic geometric mean titer (GMT) of HPV 16/18 between 6, 12, 18, and 24 months after the prime dose and prior to the administration of the second dose.

SECONDARY OBJECTIVES:

I. To determine the persistence and stability of serologic GMT of HPV types 6/11/31/33/45/52/58 between 6, 12, 18, and 24 months after prime dose and prior to the administration of the second dose.

II. To assess safety and reactogenicity to each vaccine dose.

OUTLINE:

Participants receive recombinant human papillomavirus nonavalent vaccine intramuscularly (IM) at baseline (priming injection) and at 24 and 30 months (booster injections).

After completion of study, participants are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, medically well girls and boys
* Ability to understand and the willingness to sign a written informed consent document by the legal representative(s) of the participant
* Ability to understand and the willingness to sign a written assent document by the participant

Exclusion Criteria:

* Previous vaccination against HPV
* The use of any investigational agent within 30 days preceding the first dose of the study vaccine or subsequent participation in another clinical trial at any time during the study period, in which the subject will be exposed to an investigational product
* Chronic administration of immunosuppressive agents or other immune-modifying drugs or chemotherapeutic agents within six months prior to the first vaccine dose; use of inhaled steroids, nasal sprays, and topical creams for small body areas is allowed
* Receiving active treatment for cancer or an autoimmune condition
* Confirmed or suspected immunosuppressive or immunodeficient condition
* Known bleeding disorders that preclude intramuscular injection (e.g., on anticoagulants or thrombocytopenia)
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal dysfunction, which in the opinion of the investigator precludes administration of the study vaccine
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of GARDASIL 9 (recombinant human papillomavirus nonavalent vaccine), including yeast allergy
* Are pregnant

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2026-01-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Hui (Sherry) Chow, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (2):
- United States (2):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California

REFERENCES:
- [Derived] Zeng Y, Moscicki AB, Sahasrabuddhe VV, Garcia F, Woo H, Hsu CH, Szabo E, Dimond E, Vanzzini S, Mondragon A, Butler V, DeRose H, Chow HS. A prospective, single-arm, open-label, non-randomized, phase IIa trial of a nonavalent prophylactic HPV vaccine to assess immunogenicity of a prime and deferred-booster dosing schedule among 9-11 year-old girls and boys - clinical protocol. BMC Cancer. 2019 Apr 1;19(1):290. doi: 10.1186/s12885-019-5444-4. PMID 30935375

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevention (Gardasil 9)
Started | 201
Completed | 187
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Gardasil 9)
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (0.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 131
  More than one race | 27
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 201

OUTCOME MEASURES:

1. Primary Outcome: Change in Human Papilloma Virus (HPV)16/18 Antibody Titer
Description: Difference in the log-transformed HPV 16/18 antibody levels between 6 and 12 months, between 12 and 18 months, and between 18 and 24 months after prime dose.
Time Frame: Between 6 and 24 months after prime dose and prior to the administration of the second dose
Population: Analysis on participants who provided blood samples in all study visits
Measure: Mean (Standard Deviation); unit: Log10 IU/ml
Arm/Group | Prevention (Gardasil 9)
Number analyzed (Participants) | 179
Log10 IU/ml
  Difference in HPV16 titers between 6 and 12 months | -0.55 (0.54)
  Difference in HPV16 titers between 12 and 18 months | 0.03 (0.62)
  Difference in HPV16 titers between 18 and 24 months | -0.002 (0.64)
  Difference in HPV18 titers between 6 and 12 months | -0.38 (0.46)
  Difference in HPV18 titers between 12 and 18 months | -0.005 (0.53)
  Difference in HPV18 titers between 18 and 24 months | -0.02 (0.63)

2. Secondary Outcome: Change in the Antibody Titer of Other Carcinogenic HPV Types 31/33/45/52/58 and Non-carcinogenic HPV 6/11
Description: Difference in the log-transformed HPV type-specific antibody levels between 6 and 12 months, between 12 and 18 months, and between 18 and 24 months after prime dose.
Time Frame: Data are not available. The study team is working on analyzing the antibody titers of other HPV types.
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Adverse Events, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: Up to 2 weeks post-treatment
Reporting Status: Not Posted

4. Secondary Outcome: Vaccine Reactogenicity
Time Frame: Up to 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Prevention (Gardasil 9)
All-Cause Mortality (participants affected / at risk) | 0/201
Serious Adverse Events (participants affected / at risk) | 2/201
Other Adverse Events (participants affected / at risk) | 151/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Gardasil 9) (N=201)
Appendicitis (Infections and infestations) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Gardasil 9) (N=201)
Nausea (Gastrointestinal disorders) | 13
Stomach pain (Gastrointestinal disorders) | 16
Fever (General disorders) | 11
Flu like symptoms (General disorders) | 15
Injection site reaction (General disorders) | 69
Pain (General disorders) | 11
Upper respiratory infection (Infections and infestations) | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Headache (Nervous system disorders) | 34
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT02568566/Prot_SAP_ICF_001.pdf